CLINICAL TRIAL: NCT06212947
Title: A Multicenter Multinational Observational Study of Children With Hypochondroplasia
Status: Recruiting | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 111-902
Record Dates: First submitted 2023-12-14; First posted 2024-01-19 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Hypochondroplasia
MeSH Terms: conditions — Hypochondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children with Hypochondroplasia: Children with Hypochondroplasia

SUMMARY:
This study will assess growth over time and the clinical course of HCH in children by collecting growth measurements and other variables of interest.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≤ 15 years old at the time of signing the informed consent
* Participants must have genetic confirmation of Hypochondroplasia diagnosis

Exclusion Criteria:

* Have a diagnosis of another genetic short stature condition other than Hypochondroplasia or a genetic variant known to cause another genetic syndrome associated with short stature
* Received an investigational product or medical device within 6 months before the Screening visit

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include approximately 400 pediatric individuals with hypochondroplasia.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2043-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in annualized growth velocity (AGV) | Every 6 months through end of study, up to 15 years
Change in Height Z-score | Every 6 months through end of study, up to 15 years
Change in Height | Every 6 months through end of study, up to 15 years
Change in BMI | Every 6 months through end of study, up to 15 years
Change in BMI Z-score | Every 6 months through end of study, up to 15 years
Change in ratios of upper to lower body segments | Every 6 months through end of study, up to 15 years
Change in ratios of upper and lower leg length ratio | Every 6 months through end of study, up to 15 years
Change in ratio of arms span to standing height ratio | Every 6 months through end of study, up to 15 years

SECONDARY OUTCOMES:
Change in Quality of Life in Short Statured Youth (QoLISSY) physical domain | Every 52 weeks through end of study, up to 15 years
Change in Quality of Life in Short Statured Youth (QoLISSY) total score | Every 52 weeks through end of study, up to 15 years
Change in patient global impression of severity (PGI-S) | Every 52 weeks through end of study, up to 15 years
Change in caregiver global impression of severity (CaGI-S) | Every 52 weeks through end of study, up to 15 years
Frequency of event rates of medical events of interest | Every 6 months through end of study, up to 15 years
Proportion of children who report use of growth hormone, treatment patterns and impact on growth | Every 6 months through end of study, up to 15 years
Proportion of children who report limb lengthening surgery | Every 6 months through end of study, up to 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (43):
- United States (16):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCSF Benioff Children's Hospital, Oakland, California
  - Nemours Alfred I. Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Health System, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - University of Missouri, Columbia, Missouri
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Mount Sinai Kravis Children's Hospital, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Cook Children's Endocrinology, Fort Worth, Texas
  - Medical College of Wisconsin, Children's Hospital, Milwaukee, Wisconsin
- Hospital de Pediatria SAMIC Prof. Dr. Juan P Garrahan, Buenos Aires, Argentina
- Royal Children's Hospital Melbourne, Parkville, Victoria, Australia
- Brazil (2):
  - Hospital de Clinicas de Porto Algre, Porto Alegre, Rio Grande Do Sol
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto, Ribeirão Preto, São Paulo
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - SickKids - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (4):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Lyon
  - Hopital de la Timone, Marseille
  - Hôpital Necker-Enfants Malades, Paris
  - CHU de Toulouse - Hopital des Efants, Toulouse
- Germany (2):
  - Uniklinik Koln, Cologne
  - Universitatskinderklinik Magdeburg, Magdeburg
- Italy (4):
  - Istituto Giannina Gaslini, Genoa, Liguria
  - Ospedale Pediatrico Bambino Gesù, Roma, Rome
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
- Japan (5):
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Osaka University Hospital, Suita, Osaka
  - Tottori University Hospital, Yonago, Tottori
  - Tokushima University Hospital, Tokushima
  - Institute of Science Tokyo Hospital, Tokyo
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Vithas Hospital San Jose, Vitoria-Gasteiz
- United Kingdom (3):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London, England
  - Myriad Trials Ltd, London, England
  - NHS Greater Glasgow and Clyde, Glasgow, Scottland

IPD SHARING:
Plan to Share IPD: No